CLINICAL TRIAL: NCT05812495
Title: A Multicenter,Randomized Controlled Clinical Study of Minimally Invasive Intrathoracic Esophagogastric Side to Side Anastomosis vs. End to Side Anastomosis in the Treatment of Lower Esophageal Cancer or Esophageal Gastric Junction Cancer
Brief Title: Minimally Invasive Intrathoracic Esophagogastric Side to Side Anastomosis vs. End to Side Anastomosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Peng Tang, Chief Physician, Department Director, Tianjin Medical University Cancer Institute and Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CESS2021TB01
Record Dates: First submitted 2022-12-22; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Epiphora Due to Insufficient Drainage, Left Side; Epiphora Due to Insufficient Drainage, Right Side

STUDY DESIGN:
Masking Description: Esophagogastric Side to Side Anastomosis vs. End to Side Anastomosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esophagogastric Side to Side Anastomosis (Experimental): Esophagogastric Side to Side Anastomosis
  Interventions: Procedure: Esophagogastric Side to Side Anastomosis
- Esophagogastric End to Side Anastomosis (Experimental): Esophagogastric End to Side Anastomosis
  Interventions: Procedure: Esophagogastric End to Side Anastomosis

INTERVENTIONS:
Procedure: Esophagogastric Side to Side Anastomosis — Esophagogastric Side to Side Anastomosis
  Arms: Esophagogastric Side to Side Anastomosis
Procedure: Esophagogastric End to Side Anastomosis — Esophagogastric End to Side Anastomosis
  Arms: Esophagogastric End to Side Anastomosis

SUMMARY:
On the basis of minimally invasive Ivor Lewis operation for the treatment of lower thoracic esophageal cancer or esophageal gastric junction cancer, the purpose of this study is to compare the probability of anastomotic leakage and stenosis after esophagogastric side to side anastomosis and esophagogastric end to side anastomosis, combined with the probability of complications, quality of life and survival rate of patients after the two anastomotic methods, To explore which anastomotic method is better than the worse for patients with lower thoracic esophageal cancer or cancer at the junction of esophagus and stomach. This study explored a minimally invasive anastomotic method with lower incidence of complications and higher quality of life for patients during Ivor Lewis surgery, which can increase the clinical benefits of patients, improve the quality of life, and extend the survival period, and has important clinical value.

DETAILED DESCRIPTION:
To carry out a multicenter, prospective, randomized controlled, phase III clinical study of minimally invasive Ivor Lewis operation for esophagogastric side to side anastomosis versus esophagogastric end to side anastomosis in the treatment of lower thoracic esophageal cancer or esophageal gastric junction cancer. Before grouping, introduce the similarities and differences of surgical methods to all patients, and group the patients who meet the conditions for inclusion through random control.

The specific groups are as follows:

Test group: intrathoracic esophagogastrostomy with minimally invasive Ivor Lewis operation

Control group: intrathoracic esophagogastric end-to-end anastomosis under minimally invasive Ivor Lewis operation

Each patient will be given a unique study number and will remain unchanged throughout the trial.

Main end points:

The rate of anastomotic leakage within 3 months after operation.

Secondary endpoint:

1. Incidence rate and occurrence time of anastomotic stenosis after operation;
2. Reflux esophagitis;
3. R0 resection rate, minimally invasive conversion rate, operation time, bleeding volume, number of lymph nodes cleaned, number of lymph node cleaning stations, positive rate of lymph nodes, pathological stage, chest drainage volume, drainage tube placement time, gastric tube removal time, time to start eating after operation, and hospital stay.
4. Incidence rate of intraoperative accidents
5. Incidence rate of perioperative complications (pulmonary infection, cardiovascular complications, bleeding, chylothorax, pulmonary embolism, incision infection, etc.), rate of ICU transfer, and 30 day and 90 day mortality rate;
6. Quality of life (EORTC QLQ-C30, EORTC QLQ-OES18), nutritional status score and pain score in January, March, June and year after year;
7. Patient compliance, adverse event (AE) related to treatment, incidence and severity of serious adverse events;
8. 1, 2 and 3 year Progression free survival (PFS) and Overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. The clinical staging of pathological and imaging diagnosis was cT1b-4a, N0-2, M0 stage of lower thoracic esophageal squamous cell carcinoma or Siewert type I and Siewert type II esophageal gastric junction adenocarcinoma (8th UICC-TNM staging);
2. The lesion is potentially resectable;
3. CT3-4a and/or N+patients receive neoadjuvant therapy with the informed consent of patients and their families
4. Comprehensive evaluation is suitable for Ivor Lewis operation
5. Aged 18-75 years, both male and female;
6. There was no contraindication in the preoperative examination and evaluation of various organ functions;
7. The following laboratory tests confirmed that the bone marrow, liver and kidney functions and blood coagulation met the requirements for participating in the study:

   Hemoglobin ≥ 9.0g/L;

   White blood cell count ≥ 4.0 × 109/L；

   Absolute neutrophil count (ANC) ≥ 1.5 × 109/L；

   Platelet count ≥ 100 × 109/L；

   The international standardized ratio of prothrombin time ≤ 1.5 times the upper limit of normal value, and part of the thromboplastin time is within the range of normal value;

   Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal value or creatinine clearance ≥ 50 ml/min (Cockcroft Gault formula);

   Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN);

   The level of AST or ALT ≤ 2.5 times the upper limit of normal value (ULN);

   Urine protein<2+; If the urine protein ≥ 2+, the 24-hour urine protein quantitative display must be ≤ 1g;
8. Lung function: FEV1 ≥ 1.2L, FEV1% ≥ 50% and DLCO ≥ 50%
9. Estimated lifetime ˃ 12 months.
10. R0 resection is expected;
11. The color Doppler ultrasound of the neck showed no suspicious metastatic lymph nodes;
12. Generally in good condition, individual machine energy meter (Karnofsky score, KPS) ≥ 70; Physical status ECOG 0-2 points;
13. The subjects were fully informed of the purpose of the study, voluntarily joined the study, with good compliance, safety and survival follow-up.

Exclusion Criteria:

1. Patients with cervical and upper middle thoracic esophageal cancer or Siewert III esophageal gastric junction cancer;
2. Patients with T4b stage inoperable, multiple lymph node enlargement (estimated metastasis ≥ 3), multistation lymph node enlargement (estimated lymph node metastasis ≥ 2) or distant metastasis (M1);
3. Those who can not use stomach to replace esophagus in this operation due to previous operation
4. Previous history of other malignant tumors;
5. Pathological examination of non squamous and non adenocarcinoma patients;
6. Preoperative neoadjuvant chemotherapy and radiotherapy;
7. Severe emphysema and pulmonary fibrosis;
8. Confirmed history of congestive heart failure; Angina pectoris with poorly controlled medication; Transmural myocardial infarction confirmed by electrocardiogram (ECG); Poor control of hypertension; Valvular heart disease with clinical significance; Or high risk uncontrollable arrhythmia;
9. Serious uncontrolled systemic diseases, such as active infection or poorly controlled diabetes;
10. Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg>2g/L), bleeding tendency (such as active peptic ulcer) or receiving thrombolytic or anticoagulant treatment;
11. Those who already have or are associated with hemorrhagic diseases;
12. People with peripheral nervous system disorder or obvious mental disorder and central nervous system disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of anastomotic leakage within 3 months after operation | 3 months
  The rate of anastomotic leakage within 3 months after operation

SECONDARY OUTCOMES:
Incidence rate and occurrence time of anastomotic stenosis after operation | 3 months
  Incidence rate and occurrence time of anastomotic stenosis after operation

CONTACTS AND LOCATIONS:
Overall Officials: Peng Tang, MD., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No